CLINICAL TRIAL: NCT01919996
Title: Ocular Effects Of Azithromycin Oral Solution In Pediatric Patients With Pharyngitis/Tonsillitis
Brief Title: PASS Study To Evaluate The Potential Of Zithromax To Cause Ocular Problems In Pediatric Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Termination Statement in the Detailed Description below
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661206; 208291 (Other: Alias Study Number); 2016-001119-19 (EudraCT Number)
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Pharyngitis; Tonsillitis
Keywords: Ocular safety; azithromycin; pharyngitis; tonsillitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): Azithromycin oral suspension (immediate release) 12 mg/kg/day x 5 days
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin oral suspension (immediate release) 12 mg/kg/day x 5 days

SUMMARY:
This Post-Authorization Safety Study (PASS) is intended to fulfill a regulatory post-marketing requirement to provide data regarding visual abilities in children taking azithromycin (immediate-release formulation) for acute pharyngitis/tonsillitis. The primary objective of the study is to examine the incidence of clinically significant worsening in any of the following ophthalmic exams: best corrected visual acuity (distance), color vision, Amsler grid testing, anterior segment biomicroscopy, and fundus examination, in a group of approximately 30 pediatric patients taking azithromycin oral solution for treatment of an authorized indication of use (pharyngitis/ tonsillitis).

DETAILED DESCRIPTION:
Study was terminated prematurely on October 16, 2015 following FDA decision to release Sponsor from post-marketing commitment. No safety and/or efficacy concerns identified.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, aged 12 to 17 years.
* Requires outpatient treatment for acute pharyngitis/tonsillitis infection.
* Appropriate to treat with oral azithromycin as an alternative to intramuscular penicillin, in the opinion of the investigator.
* Positive rapid antigen detection test.

Exclusion Criteria:

* History of clinically significant eye disorder that would interfere with protocol test procedures.
* Hypersensitivity to azithromycin, erythromycin, any macrolide, or ketolide antibiotic.
* Increased risk of QT prolongation.
* Pregnant or breastfeeding.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Martel Eye Medical Group, Rancho Cordova, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Outpatient Center in Lincoln Park, Chicago, Illinois
  - Infant Welfare Society of Chicago, Chicago, Illinois
  - Murray Pediatrics, Murray, Utah
  - Daynes Eye and Lasik, Salt Lake City, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661206&StudyName=PASS%20Study%20To%20Evaluate%20The%20Potential%20Of%20Zithromax%20To%20Cause%20Ocular%20Problems%20In%20Pediatric%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample size of 30 completed participants was specified by Food and Drug Administration (FDA) in the Post Marketing Commitment (PMC). Of the 30 pediatric participants planned for the study, 11 were screened and 8 participants received study treatment.
Pre-assignment Details: This was a prospective, non-comparative, open-label, single-arm study of azithromycin oral solution in 30 pediatric participants (aged 12 to 17 years) with pharyngitis/ tonsillitis who could be treated with azithromycin for their infection. The study design was intended to align with request from FDA to conduct the study.
Groups:
- Azithromycin: All participants had received open-label azithromycin oral suspension immediate release (12 mg/kg/day, up to a maximum daily dose of 500 mg) on Days 1, 2, 3, 4, and 5.
Period: Overall Study
Arm/Group | Azithromycin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants that took at least one dose of study medication.
Arm/Group | Azithromycin
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a Clinically Significant Worsening Based on Five Ophthalmic Examinations
Description: Clinically significant worsening is an observed worsening in any of the five ophthalmic exams: 1) Clinically significant worsening in best corrected visual activity (BCVA) (distance) at the final visit, in either eye, is defined as a decrease in score of 5 or more letters from baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA. 2) An assessment of abnormal clinically significant at final visit in color vision Farnsworth Munsell 100 Hue Test (FM-100) in either eye. 3) An assessment of abnormal clinically significant at final visit in Amsler Grid in either eye. 4) Assessments of abnormal clinically significant at final visit in anterior segment biomicroscopy, in any of the 10 eye structures in either eye. 5) Assessments of abnormal clinically significant at final visit in dilated indirect ophthalmoscopy in any of the 5 eye structures in either eye.
Time Frame: 14 days
Population: The safety population included all enrolled participants that took at least one dose of study medication. One participant was not evaluable because visual acuity was not corrected at Baseline (Day 1) and was corrected at Final Visit (Day 14).
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 8
percentage of participants
  Clinically significant worsening - Yes | 0.0
  Clinically significant worsening - No | 87.5
  Not Evaluable | 12.5

2. Secondary Outcome: Occurrence of a Clinically Significant Improvement Based on Five Ophthalmic Examinations
Description: 1 or more of these conditions are clinically significant improvement based on five ophthalmic exams:1) clinically significant improvement in BCVA(distance) at the final visit, in either eye, defined as an increase in score of 5 or more letters from baseline in ETDRS BCVA.2) Assessment of abnormal clinically significant at baseline and normal or abnormal, non-clinically significant at final visit in color vision(FM-100) in either eye. 3) Assessment of abnormal clinically significant at baseline and normal/abnormal, non-clinically significant at final visit in Amsler Grid in either eye. 4) Assessments of abnormal clinically significant at baseline and normal/abnormal, non-clinically significant at final visit in anterior segment biomicroscopy, in any of the 10 eye structures in either eye. 5)Assessments of abnormal clinically significant at baseline and normal/abnormal, nonclinically significant at final visit in dilated ophthalmoscopy in any of the 5 eye structures in either eye.
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 8
percentage of participants
  Clinically Significant Improvement - Yes | 12.5
  Clinically Significant Improvement - No | 75.0
  Not Evaluable | 12.5

3. Secondary Outcome: Occurrence of a Clinically Significant Change (Improvement or Worsening) Based on Five Ophthalmic Examinations
Description: Clinically significant change (improvement or worsening) is based on five ophthalmic exams at baseline and the final visit. Any 1 or more of these conditions are a clinically significant change: 1) A worsening in BCVA (distance), as defined in outcome measure 1 OR an improvement in BCVA (distance) as defined in outcome measure 2. 2) A worsening in color vision (FM-100), as defined in outcome measure 1 OR an improvement in color vision (FM-100) as defined in outcome measure 2. 3) A worsening in Amsler Grid, as defined in outcome measure 1, OR an improvement in Amsler Grid, as defined in outcome measure 2. 4) A worsening in anterior segment biomicroscopy, as defined in outcome measure 1 OR an improvement in anterior segment biomicroscopy as defined in outcome measure 2. 5) A worsening in dilated indirect ophthalmoscopy, as defined in outcome measure 1 OR an improvement in dilated indirect ophthalmoscopy as defined in outcome measure 2.
Time Frame: 14 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 8
percentage of participants
  Significant Change (Improvement or Worsening) -Yes | 12.5
  Significant Change (Improvement or Worsening) - No | 75.0
  Not Evaluable | 12.5

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 calendar days after the last administration of the study medication (up to 40 days)
Description: The safety population included all enrolled participants that took at least one dose of study medication.
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
The study was terminated after the FDA released the Sponsor from the PMC. The FDA deemed the study as impracticable, given the azithromycin dose studied in the PMC was not used and the available data did not identify a signal for ocular toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.